CLINICAL TRIAL: NCT06243770
Title: A Phase 1, Randomized, Open-label, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-0184 Administered Under Different Infusion Conditions in Healthy Participants
Brief Title: Study to Investigate Safety and Tolerability of mRNA-0184 Administered Under Different Infusion Conditions in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: mRNA-CRTX-001
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: mRNA-0184; Messenger RNA; Moderna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort 1: mRNA-0184 Dose Level A (Experimental): Sequence 1: Participants will receive infusion condition 1 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 2 of mRNA-0184 on Day 22.
  Sequence 2: Participants will receive infusion condition 2 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 1 of mRNA-0184 on Day 22.
  Interventions: Drug: mRNA-0184
- Cohort 2: mRNA-0184 Dose Level B (Experimental): Sequence 1: Participants will receive infusion condition 1 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 2 of mRNA-0184 on Day 22.
  Sequence 2: Participants will receive infusion condition 2 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 1 of mRNA-0184 on Day 22.
  Interventions: Drug: mRNA-0184
- Cohort 3: mRNA-0184 Dose Level C (Experimental): Sequence 1: Participants will receive infusion condition 1 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 2 of mRNA-0184 on Day 22.
  Sequence 2: Participants will receive infusion condition 2 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 1 of mRNA-0184 on Day 22.
  Interventions: Drug: mRNA-0184
- Cohort 4: mRNA-0184 Dose Level D (Experimental): Sequence 1: Participants will receive infusion condition 3 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 4 of mRNA-0184 on Day 22.
  Sequence 2: Participants will receive infusion condition 4 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 3 of mRNA-0184 on Day 22.
  Interventions: Drug: mRNA-0184
- Cohort 5: mRNA-0184 Dose Level E (Experimental): Sequence 1: Participants will receive infusion condition 5 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 6 of mRNA-0184 on Day 22.
  Sequence 2: Participants will receive infusion condition 6 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 5 of mRNA-0184 on Day 22.
  Interventions: Drug: mRNA-0184
- Cohort 6: mRNA-0184 Dose Level F (Experimental): Sequence 1: Participants will receive infusion condition 5 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 6 of mRNA-0184 on Day 22.
  Sequence 2: Participants will receive infusion condition 6 of mRNA-0184 on Day 1, followed by a washout period of approximately 21 days. They will then receive infusion condition 5 of mRNA-0184 on Day 22.
  Interventions: Drug: mRNA-0184

INTERVENTIONS:
Drug: mRNA-0184 — Intravenous infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of intravenously (IV) administered mRNA-0184 under different infusion conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, electrocardiogram (ECG), and vital signs.
2. Participant who could become pregnant must meet conditions as defined in the protocol.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
2. Any clinically significant illness, or medical/surgical procedure, within 4 weeks of the first administration of the study investigational product (IP) (mRNA-0184).
3. Any clinically significant abnormalities in clinical laboratory results at Screening. Repeat assessments are allowed at the Investigator's discretion if a false positive is suspected.
4. Clinically significant abnormal findings in vital signs at Screening.
5. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
6. Use of any prescribed medication during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of the study IP. Hormonal contraception is permitted.
7. Has received another IP within 4 weeks of the first dosing of the study IP or within 5 terminal half-lives of the IP, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 57
Number of Participants with Adverse Events of Special Interest (AESIs) | Day 1 through Day 57
Number of Participants with Serious Adverse Events (SAEs) | Day 1 through Day 57

SECONDARY OUTCOMES:
Serum Concentrations of Study Drug | Day 1 through Day 57
Maximum Concentration (Cmax) of Study Drug | Day 1 through Day 57
Area Under the Concentration-time Curve from Time 0 to Last Quantifiable Concentration (AUC0-t) of Study Drug | Day 1 through Day 57
Serum Concentrations of Relaxin-2-variable Light Chain Kappa (Rel2- vlk) Protein | Day 1 through Day 57
Maximum Observed Response (Emax) of Rel2- vlk Protein | Day 1 through Day 57
Area Under the Effect-time Curve (AUEC) of Rel2- vlk Protein | Day 1 through Day 57
Number of Participants with Anti-Polyethylene Glycol (PEG) Antibodies | Day 1 through Day 57
Number of Participants with Anti-Rel2-vlk Protein Antibodies | Day 1 through Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia